CLINICAL TRIAL: NCT02355600
Title: Tamoxifen as Adjuvant Treatment in Breast Cancer and Its Impact on Ovarian Function
Brief Title: Oocyte Recovery During Tamoxifen Adjuvant Therapy
Acronym: TAMOXIFERT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/0642
Record Dates: First submitted 2015-01-22; First posted 2015-02-04 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: Oocyte; Tamoxifen; Fertility preservation
MeSH Terms: conditions — Breast Neoplasms | interventions — Oocyte Retrieval

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Oocyte retrieval — Tamoxifen given at a fixed dose for invasive breast cancer adjuvant hormonotherapy or for breast cancer prophylaxis.
  Other Names: Oocyte pick-up

SUMMARY:
Survival in young patients with cancer has increased and also have increased the adverse long-term side effects of chemotherapy, there is a large number of women who experience loss of ovarian function without accomplishing their reproductive desire due to gonadotoxic treatment. The ovarian reserve determine the response to controlled ovarian hyperstimulation in fertility preservation treatments as well as in assisted reproduction techniques. Improving this reserve by avoiding its depletion during the process could result in increase fertility rates after cancer treatment.

Collecting follicles during tamoxifen treatment would increase the number of cryopreserved oocytes and thus rise the potential ovarian reserve in these patients, which is reduced due to age, chemotherapy and length of treatments.

The aim of this study is to retrieve viable mature oocytes during adjuvancy with tamoxifen in breast cancer patients to improve the probability of subsequent pregnancy.

DETAILED DESCRIPTION:
New chemotherapy regimens and management options developed during the last 20 years have yielded increased survival rates in cancer patients but they also cause side effects such as premature ovarian failure and infertility due to their gonadotoxicity. Hormone therapy also increases survival rates in breast cancer patients; tamoxifen, a selective estrogen receptor modulator, has been proven to reduce the risk of recurrence and mortality due to breast cancer when administered during 10 years.

The risk of premature ovarian failure depends not only on the gonadotoxicity of chemotherapy but also on the age of the patient, therefore although tamoxifen is not gonadotoxic itself, it can compromise fertility because of the long length of treatment and the subsequent delay in childbearing.

On the other hand, tamoxifen is a drug that can be used in assisted reproduction techniques to induce ovarian stimulation, therefore, the tamoxifen treatment followed by breast cancer patients represent somehow a way of continuous ovarian stimulation. If viable oocytes could be retrieved during the long-term hormonal treatment with tamoxifen, there will be an option to use them to restore fertility afterwards.

STUDY DESIGN:

Patients included in the study who have normal menstrual periods will be monitored by sonography (antral follicle count) and serum hormonal levels: E2 (oestradiol), P4 (progesterone), FSH (follicle stimulating hormone) and LH (luteinizing hormone) from the second day of their cycle. Patients without spontaneous menstruations will perform periodic visits every 15 days until images corresponding with antral follicle definition will be seen, this will be considered day 2 of the cycle.

Follow-up of the antral follicles will be done with sonography and serum hormonal levels according to the protocols of the investigators in vitro fertilization unit. When a follicle of more than 18 mm is seen, 250 µg of hCG (human chorionic gonadotropin) will be administered and 36 hours after, transvaginal oocyte retrieval will be performed. Oocyte and embryo quality assessment will be performed according to morphological ASEBIR (association for the study of reproduction biology) classification on day +2 and +3. Grade 1 and 2 embryos on day +3 will be cryopreserved.

Patients requiring assisted reproduction technologies to get pregnant after completion of their oncologic treatment will have their embryos thawed and subsequently transferred.

FOLLOW-UP:

During the time oocytes retrieved are being used or until the end of gestation in case the patient become pregnant.

Bearing in mind that most of the patients in our center undergo 5 year of tamoxifen treatment, it will be assumed a maximum follow-up of 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients whose tumors have positive hormone receptors (ER+) subsidiary of adjuvant treatment with tamoxifen
* Reproductive desire

Exclusion Criteria:

* Having received chemotherapy agents less than 12 months ago
* Current treatment with GnRH analogues
* Age > 35 years old
* Contraindication for follicular punction or hCG administration

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young breast cancer patients (with positive estrogen receptors) using tamoxifen as adjuvant treatment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-11; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Metaphase II oocytes retrieved | 24 months

SECONDARY OUTCOMES:
Number of frozen embryos | 24 months
Morphologic score of frozen embryos | 24 months
Pregnancy rate | Expected average of 6 years
  pregnancy rates after the use of frozen embryos generated during tamoxifen treatment

CONTACTS AND LOCATIONS:
Overall Officials: César Diaz-Garcia, MD, Principal Investigator — IIS La Fe
Locations (1):
- Hospital Universitari i Politècnic La Fe, Valencia, Valencia, Spain